CLINICAL TRIAL: NCT06512311
Title: Personalized Targeted Glioblastoma Therapies by ex Vivo Drug Screening: Advanced Brain Tumor TheRApy Clinical Trial (ATTRACT)
Brief Title: Personalized Targeted Glioblastoma Therapies by ex Vivo Drug Screening
Acronym: ATTRACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Anna Berghoff, Assoc.-Prof. PD DDr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ATTRACT
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDC-based drug screening (Experimental): 120 patients will be included in the intervention group and will receive PDC-based drug screening. The molecular tumor board will formulate a personalized treatment recommendation by incorporating the individual characteristics of the patients including age, co-morbidities, co-medication, and performance status in addition to the results of the PDC-based drug screening.
  Interventions: Diagnostic Test: CBMed Drug Screening Plattform
- Standard group (No Intervention): 120 patients will be included in the standard group and will not receive PDC-based drug screening. In line, no personalized treatment approach will be formulated by the molecular tumor board and patients will all receive the recommendation for standard treatment including temozolomide maintenance therapy for 6 cycles.

INTERVENTIONS:
Diagnostic Test: CBMed Drug Screening Plattform — The main devices used within the drug screening process are purchased from PerkinElmer, Liconic Instruments, BioTek and Beckman Coulter Diagnostics.
  Arms: PDC-based drug screening

SUMMARY:
Patient derived cell line (PDC) -based drug screening will be applied to formulate a personalized treatment approach.

DETAILED DESCRIPTION:
Patient derived cell line (PDC) -based drug screening will be applied to formulate a personalized treatment approach. Patients will be randomized between the investigational group receiving in addition to standard histology analysis also the PDC-based drug screening and the standard group receiving only standard histology analysis. Outcome results will be compared in a randomized, interventional clinical performance study. The PDC-based drug screening will be performed only in accordance with the approved Performance Study Plan on subjects who have signed an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* ECOG performance status 0-2
* Newly diagnosed glioblastoma, IDH wildtype - according to the 2021 WHO classification of Tumors of the Central Nervous System
* MGMT promotor unmethylated per local investigator
* Tissue available for drug screening (successful PDC establishment from surgical material)
* Scheduled for concomitant radio-chemotherapy with temozolomide
* Written informed consent

Exclusion Criteria:

* Current participation in another therapeutic clinical trial
* Patients with a concurrent malignancy or malignancy within five years prior of study enrolment except for carcinoma in situ of the cervix, non-melanoma skin carcinoma or stage I uterine cancer within the last 3 years
* Pregnant or lactating women
* Current known infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antibody [HBsAg] test and a positive anti-hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for anti-HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Known human immunodeficiency virus (HIV) infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA, CD4+ count ≥350 cells/mm3 , no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen). If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended.
* Any of the following co-morbidities:

  * Pre-existing severe peripheral neuropathy (> CTCAE grade 2)
  * Hepatic impairment (Bilirubin Level >1.5x-3x ULN)
  * Kidney dysfunction (CrCl < 59 mL/min)
  * Cardiac dysfunction with left ventricular ejection fraction <60 %
  * Any grade of interstitial lung disease
  * Ongoing or previous history of rhabdomyolysis
  * Acute pancreatitis
  * QTcF ≥480 msec
  * Diabetes mellitus with fasting glucose > 250mg/dl or 13.9 mmol/L
* Participants who are unable or unwilling to comply with the requirements of the protocol as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | From date of randomization until date of death from any cause or last follow up whichever came first, assessed up to 144 months
  Change in overall survival in patients receiving extensive diagnostic work up including the standard histology analysis and PDC- based drug screening in addition (interventional arm) compared to patients receiving only standard histology diagnostic work up (standard arm)

SECONDARY OUTCOMES:
Feasibility of PDC-based drug screening | From date of randomization until date of communication of the tumor board outcome, asses up to 144 months
  Number not interpretable results of the PDC-based drug screening; Number of interpretable results of the PDC-based drug screening
Comparison of Quality of life measurements | From date of randomization until date of death from any cause or last follow up whichever came first, assessed up to 144 months
  Difference between the interventional and the standard arm using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ- C30) and the brain cancer specific questionnaire (QLQ-BN20). The scale is from 0 to 100, with higher values reporting better quality of life.
Comparison of neurocognitive function scale | From date of randomization until date of death from any cause or last follow up whichever came first, assessed up to 144 months
  differences in neurocognitive function between the interventional and standard arms using the Neurologic Assessment in Neuro-Oncology (NANO) scale

CONTACTS AND LOCATIONS:
Locations (1):
- AKH Vienna, Department for Internal Medicine I, Oncology, Vienna, Austria

REFERENCES:
- [Derived] Berghoff AS, Mair MJ, Spiro Z, Abdel Malak C, El-Heliebi A, Eckert F, Furtner J, Konig F, Leibetseder A, Nowosielski M, Oberndorfer S, Prietl B, Pichler J, Pieber TR, Spiegl-Kreinecker S, Urbanic Purkart T, Wohrer A, Widhalm G, Preusser M; ATTRACT study group. Personalized targeted glioblastoma therapies by ex vivo drug screening: Study protocol of the Advanced brain Tumor TheRApy Clinical Trial (ATTRACT). Neurooncol Adv. 2025 Mar 7;7(1):vdaf056. doi: 10.1093/noajnl/vdaf056. eCollection 2025 Jan-Dec. PMID 40351832